CLINICAL TRIAL: NCT05066906
Title: Assessing Videogame-Based Tool for Job Search and Executive Function Improvement in Adults With Autism Spectrum Disorder
Brief Title: Videogame-based Tool for Job Search and Executive Function Improvement in Adults With ASD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in lab priority
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Lawrence Fung, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-52313
Record Dates: First submitted 2021-05-06; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Randomization into two groups A and B. Group Intervention or group A will comprise of participants who will be given usual referrals to pre-employment training, and will not use Identifor or Companion app. Intervention or group B will comprise of participants who were randomly selected to use Identifor and Companion app, in addition to referrals to pre-employment training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of Identifor and Companion+referral to employment agencies (Experimental): This group will use the Identifor tool and Companion app for a period of 6 months. They will also receive standard referral to employment agencies.
  Interventions: Device: Use of Identifor assessment tool and Companion app; Other: Referral to employment agencies
- Referral to employment agencies (Active Comparator): This group will not use the Identifor tool and Companion app. They will only receive standard referral to employment agencies.
  Interventions: Other: Referral to employment agencies

INTERVENTIONS:
Device: Use of Identifor assessment tool and Companion app — Identifor pinpoints what players excel at by using objective metrics and quantifiable data to collect information relevant to employment, including Multiple Intelligence, Executive Function, and personality themes.
  Companion is a 24/7 personalized aide for teens and adults iwth special needs that uses and artificial intelligence avatar to have back-and-forth conversations with users in a meaningful way to support the user in different domains of their everyday lives including public transit, managing personal schedules, and money management.
  Arms: Use of Identifor and Companion+referral to employment agencies
Other: Referral to employment agencies — Standard referral to employment agencies based on an individual's background, skillset, and preferences

SUMMARY:
This study aims to assess the efficacy of Identifor, a strength- based, person-centered, vocational assessment tool to develop a more effective way to identify individual abilities, skills, and interests. Identifor uses computer games specifically designed for young adults with ASD.

ELIGIBILITY:
Inclusion Criteria:

* IQ above 60
* Diagnosis of ASD as confirmed by qualified clinician (including Dr. Fung), and if necessary the administration of Autism Diagnostic Interview-Revised (ADI-R) and/or Autism Diagnostic Observation Schedule-Generic (ADOS-G)
* Age 18 to 55
* Adults who are physically healthy
* able to travel to work independently

Exclusion Criteria:

* DSM-5 diagnosis of other severe psychiatric disorder such as schizophrenia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Rate of securing internship, part-time, or full-time positions | 6 months after initiation of referral
  Percentage of participants securing internship, part-time, or full-time positions
Level of satisfaction | 3 months after initiation of referral
  The level of participant satisfaction will be determined from a Likert scale ("Very satisfied", "Somewhat satisfied", "Neither satisfied nor dissatisfied", "Somewhat dissatisfied", and "Very dissatisfied").

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function for Adults (BRIEF-A) | 6 months after initiation of referral
  measure of executive function for adults

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fung, MD,PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No